CLINICAL TRIAL: NCT02559856
Title: Comparison of Bleeding Risk Between Rivaroxaban and Apixaban for the Treatment of Acute Venous Thromboembolism: The Pilot Study
Brief Title: Comparison of Bleeding Risk Between Rivaroxaban and Apixaban: The Pilot Study
Acronym: COBRRA Pilot
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Venous Thromboembolism Clinical Trials and Outcomes Research (CanVECTOR) Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COBRRA Pilot; 20150574-01H (Other: OHSN REB)
Record Dates: First submitted 2015-09-21; First posted 2015-09-24 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — apixaban; Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apixaban (Active Comparator): 10 mg PO twice-a-day for 1 week, then 5 mg PO, twice daily for 3 or 6 months of treatment.
  Interventions: Drug: Apixaban
- Rivaroxaban (Active Comparator): 15 mg PO twice-a-day for 3 weeks, then 20 mg PO once daily for 3 or 6 months of treatment.
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Apixaban
  Other Names: Eliquis
  Arms: Apixaban
Drug: Rivaroxaban
  Other Names: Xarelto
  Arms: Rivaroxaban

SUMMARY:
This vanguard pilot study compares rivaroxaban and apixaban, two of the new oral blood thinners for the treatment of blood clots. Half of the patients will receive apixaban and half will receive rivaroxaban. The main objective is to determine the feasibility of patient recruitment and resources required to follow enrolled patients and inform for a larger, multi-centered trial and to assess which one is safer.

DETAILED DESCRIPTION:
Recently developed new oral anticoagulants (OAC) overcome some of the limitations of established therapy with vitamin K antagonists (VKA) and low molecular weight heparin (LMWH) for treatment of acute venous thromboembolism (VTE), due to ease of administration and more predictable pharmacokinetic properties. Many clinical questions about the new OAC remain unanswered because there have not been direct head-to-head comparison trials. For example, although studies have shown that rivaroxaban and apixaban are at least as effective and safe as LMWH and VKA, meta-analyses suggest that apixaban may be associated with lower bleeding risk. Concerns about the potential impact of medication non-adherence have been raised. Compliance with twice daily medications (e.g. apixaban) is often worse than once daily medications (e.g. rivaroxaban). Both of these medications are approved by Health Canada for treatment of VTE yet there is genuine uncertainty about which of the two direct OAC confer the best risk-to-benefit ratio.This is a multi-centre, prospective randomized open blinded end-point (PROBE) trial assessing clinical feasibility for a larger multi-centered trial comparing bleeding outcomes using apixaban vs. rivaroxaban for treatment of acute VTE. The primary objective of the study is to determine if it is feasible to conduct a large randomized multicenter trial comparing apixaban vs. rivaroxaban for the treatment of acute VTE. The secondary objectives are to assess safety and superiority of apixaban vs rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed newly diagnosed acute VTE (proximal lower extremity deep vein thrombosis and segmental or greater pulmonary embolism)
* Age ≥ 18 years old
* Written informed consent

Exclusion Criteria:

* Any contraindication for anticoagulation such as active bleeding
* Clinically significant liver disease or alanine aminotransferase (ALT) levels ≥ 3 times the upper limit of normal range
* Creatinine clearance < 30 ml/min calculated with the Cockcroft-Gault formula (29)
* Known allergies to either apixaban or rivaroxaban
* Pregnancy
* Use of contraindicated medications with apixaban or rivaroxaban
* Active malignancy in the last 6 months (excluding localized skin malignancy)
* No private insurance coverage for the study drug or not willing to pay for study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients screened who are eligible to participate in the trial | For the duration of the study 3-6 months
  Assessing clinical feasibility for a larger multi-center trial - number of screened patients versus eligible patients
Proportion of eligible patients who consent to participate in the trial | For the duration of the study 3-6 months
  Assessing clinical feasibility for a larger multi-center trial - number of eligible patients versus patients who consent to participate
Proportion of patients who attend each follow-up visit | For the duration of the study 3-6 months
  Assessing clinical feasibility for a larger multi-center trial - number of patients that miss visits versus patients that attend visits.
Proportion of patients completing all required study procedures, per follow-up visit | For the duration of the study 3-6 months
  Assessing clinical feasibility for a larger multi-center trial - number of patients that complete all required procedures/study visits versus patients that do not.

SECONDARY OUTCOMES:
Bleeding Events | For the duration of the study 3-6 months
  Major bleeding events, clinically relevant non-major and minor bleeding episodes
Venous Thromboembolism | For the duration of the study 3-6 months
  Recurrent VTE and VTE related-death
Death | For the duration of the study 3-6 months
  * All-cause mortality rates
  * Individual rates of death related to VTE, cardiovascular disease, bleeding or other causes
Medication compliance | For the duration of the study 3-6 months
  As assessed by study pill count
Time-to-event analysis | For the duration of the study 3-6 months
  The time-to-first occurrence of secondary outcomes between randomization and end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lana Castellucci, MD, FRCPC, Principal Investigator — Ottawa Hospital Research Institute
Locations (4):
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - Hamilton General Hospital, Hamilton, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Hôtel-Dieu de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No